CLINICAL TRIAL: NCT06537947
Title: A Single Center, First in Human Study to Evaluate the Feasibility of the SENTANTE Robotic System Application in Peripheral Endovascular Interventions
Brief Title: SENTANTE: Fully Robotic Peripheral Endovascular Interventions
Acronym: ESSENTIAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inovatyvi Medicina UAB (Industry)
Collaborators: KCRI (Other); SIA Kotello (Unknown); Syntropic Corelab (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 24-SEN-002; CIV-24-05-047118 (Other: EUDAMED)
Record Dates: First submitted 2024-07-29; First posted 2024-08-05 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Any Disease Which Requires Peripheral Endovascular Intervention
Keywords: robotic; endovascular; SENTANTE; robot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (1):
- Endovascular interventions (Experimental)
  Interventions: Procedure: Endovascular intervention using the SENTANTE endovascular robotic system

INTERVENTIONS:
Procedure: Endovascular intervention using the SENTANTE endovascular robotic system — 1. Diagnostic procedure - placement of diagnostic catheter to intended vessel and performing angiography.
  2. Percutaneous transluminal angioplasty (PTA)/stenting procedure - placement of balloon catheter or balloon expandable stent to intended vessel and effectively expanding it up to nominal pressure.
  3. Coiling procedure - implantation of pushable coils or liquid embolization materials (such as microspheres) to an intended vessel.

SUMMARY:
The objective of the study is to evaluate the feasibility, safety and initial efficacy of the clinical and technical performance of the SENTANTE robotic system in the remote delivery and manipulation of commonly used and compatible guidewires and catheter-based devices for use in peripheral endovascular procedures.

The study will be a single-center, prospective investigation, designed to evaluate the safety, feasibility, and initial efficacy of robotic system for remote endovascular interventions in adults with disease which requires peripheral endovascular treatment with compatible devices. Participants meeting the inclusion criteria will undergo endovascular interventions using SENTANTE robotic system. Data will be collected through clinical assessments, imaging and other studies, laboratory tests, and feedback from medical personnel and patients.

The study will adhere to ethical guidelines, obtain informed consent from all participants, and be conducted under the oversight of the Clinical Events Committee.

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≥ 19 years and ≤ 90 years of age.
* Subject is willing and able to provide appropriate study-specific informed consent and follow Clinical Investigation Plan (CIP) procedures.
* Life expectancy ≥ 12 months from the date of the index procedure.
* Females who are not pregnant or lactating and not planning to become pregnant for the duration of the study.
* Subject is diagnosed with a disease which requires peripheral endovascular intervention using compatible with SENTANTE guidewires and catheter-based devices.

Exclusion Criteria:

* Planned interventional procedure or surgery of the carotid, coronary or peripheral arteries within 30 days before or after the index procedure.
* Subjects with myocardial infarct or cerebrovascular event within 3 months prior to index procedure.
* Severe vascular anatomy that would preclude safe sheath insertion, or deliverability of stent.
* History of bleeding diathesis or coagulopathy.
* History of thrombophilia.
* Sensitivity to contrast media that cannot be adequately pre-treated.
* Sensitivity to both forms of CIP-acceptable anticoagulation strategies (i.e., both heparin AND Bivalirudin).
* Sensitivity to an antiplatelet agent AND all CIP acceptable alternative antiplatelet options.
* Major neurologic deficit with NIHSS of ≥ 15.
* Clinical condition that, in the opinion of the investigator, makes endovascular therapy impossible or hazardous.
* Subject previously enrolled in this clinical trial.
* Possible / probable non-compliance of subject with CIP required follow up or medication.
* Subject is currently participating in another clinical trial that has not completed its primary endpoint assessment or would confound this Clinical Study.
* Signs of SARS-CoV2 (COVID-19) active infection.
* Patients with intervention-related anxiety, separation anxiety, autophobia and individuals that cannot be left alone without additional sedation or close supervision.

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2024-07-19 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Efficacy endpoint: Number of procedures with technical success | Immediately after intervention
  Technical success rate counted per procedure basis, defined as:
  i. Diagnostic procedure - placement of diagnostic catheter to intended vessel and performing angiography.
  ii. PTA/stenting procedure - placement of balloon catheter or balloon expandable stent to intended vessel and effectively expanding it up to nominal pressure.
  iii. Coiling procedure - implantation of pushable coils or liquid embolization materials (such as microspheres) to an intended vessel.
Safety endpoint: Number of procedures without adverse device effects (ADEs) | Immediately after intervention and after 96 hours post procedure or hospital discharge if comes first
  Safety level counted per procedure basis, defined as absence of evidence of device related clinically significant vessel injury, with particular emphasis on events such as:
  i. Perforation, ii. Thrombosis, iii. Flow limiting residual dissection, iv. Distal embolization (excluding embolization procedure). The assessment of the impact of observed ADEs on the safety profile of the robotic system will be based on the Clinical event committee (CEC) adjudication.

SECONDARY OUTCOMES:
Procedural success: Number of procedures with achieved success | Immediately after intervention and after 96 hours post procedure or hospital discharge if it comes first
  Procedure success is defined depending on the type of procedure as follows:
  i. Diagnostic procedure - sufficient diagnostic information was achieved to make further decisions on treatment plan.
  ii. Treatment of stenotic lesions / occlusions - <50% residual stenosis in all SENTANTETM Robotic System treated lesions at the completion of the interventional procedure without an unplanned switch to the manual procedure in the absence of ADEs.
  iii. Treatment of bleeding or other diseases requiring embolization - successful occlusion of SENTANTETM robotic system treated vessels at the completion of the interventional procedure without an unplanned switch to the manual procedure in the absence of ADEs.
Rate of manual assistance | During the intervention
  Device manipulation requiring manual assistance during fluoroscopy, evaluated per procedure
Rate of conversion to manual procedure | During the intervention
  Performance of procedural steps manually instead of manipulation with a robotic system
Successful advancement/retrieval of the device without manual assistance | During the intervention
  The manipulation (advancement/retrieval) of endovascular devices with the SENTANTE robotic system will be evaluated per device basis
Clinical success | Immediately after intervention and after 96 hours post procedure or hospital discharge if comes first
  Number of patients with confirmation that the performed intervention has achieved its intended therapeutic effect or clinical benefit
Safety level at access site | After 96 hours post procedure or before hospital discharge if it comes first
  Number of patients without adverse events
Radiation exposure in a typical operator workplace | Immediately after intervention
  Amount of radiation exposure while using robotic system
Procedural satisfaction reported by patients on dedicated form | Within 96 hours post procedure or before hospital discharge if it comes first
  Questionnaire to be completed by the patient after the intervention. Questionnaire consists of 8 questions. The response to each question is asked to be evaluated on a scale from 1 to 4, with 1 representing the favorable aspect of the characteristic described in the question and 4 representing the least favorable aspect of the characteristic described in the question.
Operator feedback on dedicated form | Within 96 hours post procedure
  Questionnaire to be completed by the Operator after the intervention. Questionnaire consists of 10 questions. The response to each question is asked to be evaluated on a scale from 1 to 4, with 1 representing the favorable aspect of the characteristic described in the question and 4 representing the least favorable aspect of the characteristic described in the question.
Nurse feedback on dedicated form | Within 96 hours post procedure
  Questionnaire to be completed by the assisting personnel after the intervention.
  Questionnaire consists of 8 questions. The response to each question is asked to be evaluated on a scale from 1 to 4, with 1 representing the favorable aspect of the characteristic described in the question and 4 representing the least favorable aspect of the characteristic described in the question.
Clinical events (adverse event (AE)/serious adverse event (SAE)/adverse device effect (ADE)) during the index procedure and till the discharge | Immediately after intervention and within 96 hours post procedure or before hospital discharge if it comes first
  Recorded and reported clinical events

CONTACTS AND LOCATIONS:
Overall Officials: Dainis Krievins, Prof PhD MD, Principal Investigator — Pauls Stradins Clinical University Hospital
Locations (1):
- Pauls Stradins Clinical university hospital, Riga, Latvia